CLINICAL TRIAL: NCT01272466
Title: Vaccination With Peptides Derived From Anti-apoptotic Proteins From the Bcl-2 Family, Administered in Combination With Montanide ISA-51 in Relation to Treatment With Proteasome Inhibitors in Patients With Relapsed Multiple Myeloma
Brief Title: Vaccination With Peptides From Anti-apoptotic Proteins in Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lene Meldgaard Knudsen, M.D, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-003619-29
Record Dates: First submitted 2011-01-03; First posted 2011-01-07 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Relapsed Multiple Myeloma
Keywords: multiple myeloma; vaccination; antiapoptotic proteins; proteasome inhibition
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- peptides from antiapoptotic proteins (Experimental)
  Interventions: Biological: peptides derived from antiapoptotic proteins

INTERVENTIONS:
Biological: peptides derived from antiapoptotic proteins — 8 Vaccinations on day 2 and 9 in every bortezomib treatment series

SUMMARY:
Anti-apoptotic proteins from the Bcl-2 family are known to play a key role in oncogenesis and are overexpressed in myeloma cells. Studies have shown that dendritic cells exposed to proteasome inhibition present exogene antigens better than unexposed dendritic cells. Patients with relapse of multiple myeloma will be offered vaccination with peptides derived from antiapoptotic proteins from the Bcl-2 family in combination with an immunostimulatory adjuvant. The vaccination will be given in relation to treatment with the proteasome inhibitor bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of multiple myeloma
* tissue type of HLA-A1, HLA-A2 or HLA-A3
* Performance status < 2
* Adequate bone marrow - renal and liver function
* written informed concent

Exclusion Criteria:

* candidate for bone marrow transplantation
* other malignancies than multiple myeloma
* other significant medical disease (heart-, lung or liver disease or diabetes)
* allergy
* active autoimmune disease
* treatment with immunosuppressive drugs
* treatment with other experimental drugs
* uncontrolled hypercalcemia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Lene M Knudsen, M.D, Principal Investigator — Department of Haematology, Odense University Hospital
Locations (1):
- Department of Haematology, Odense University Hospital, Odense, Denmark